CLINICAL TRIAL: NCT03432208
Title: A Pilot Study to Assess the Potential Value of Adding Endoscopic Ultrasound (EUS) to Esophago-gastro-duodenoscopy (EGD) in Emergency Room Patients Referred for Egd
Brief Title: A Pilot Study to Assess the Value of EUS vs EGD in Emergency Room Patients Referred for EGD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by CHUM REB for lack of documentation related to the recruitment of participants.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, A Sahai, Professeur Adjoint, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 14.320
Record Dates: First submitted 2016-05-11; First posted 2018-02-14 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESOPHAGO-GASTRO-DUODENOSCOPY (EGD) (Active Comparator): GI consult Procedure performed is EGD
  Interventions: Procedure: GI consult
- ENDOSCOPIC ULTRASOUND (EUS) (Experimental): GI consult Procedure performed is EUS
  Interventions: Procedure: GI consult

INTERVENTIONS:
Procedure: GI consult

SUMMARY:
Emergency room patients referred for esophago-gastro-duodenoscopy (EGD) often have many possible causes for their symptoms. These inevitably undergo further testing if EGD is inconclusive, which adds costs and inevitably prolongs emergency room length of stay (LOS).EUS has traditionally been used after EGD for a myriad of costs reasons that no longer apply. We therefore propose a prospective pilot study to determine whether PEUS can reduce LOS and resource utilisation in emergency room patients referred for EGD.

DETAILED DESCRIPTION:
A PILOT STUDY TO ASSESS THE POTENTIAL VALUE OF ADDING ENDOSCOPIC ULTRASOUND (EUS) TO ESOPHAGO-GASTRO-DUODENOSCOPY (EGD) IN EMERGENCY ROOM PATIENTS REFERRED FOR EGD

P.I.: Anand V. Sahai MD, MSc (EPID), FRCPC

BACKGROUND Emergency room patients referred for esophago-gastro-duodenoscopy (EGD) often have many possible causes for their symptoms. These inevitably undergo further testing if EGD is inconclusive, which adds costs and inevitably prolongs emergency room length of stay (LOS).

Endoscopic ultrasound (EUS) combines EGD with high-resolution ultrasound imaging of pancreas, liver and biliary system and is the best test to diagnose bile duct stones, early chronic pancreatitis, and small [<2cm] pancreatic cancers (all of which cannot be seen by regular ultrasound or CT scanning or MRI, yet are included in the differential diagnosis of EGD-negative abdominal pain).

EUS has traditionally been used after EGD, due to lack of availability, increased cost, and to increased risk due to larger scope diameter. However, the latest generation of EUS scopes have the same outer diameter as conventional gastroscopes, there is much wider availability of EUS in university and community hospital settings, and the cost per procedure is lower, due to increased procedural numbers and reduced maintenance costs.

In experienced hands, diagnostic EUS is now as safe and as EGD accurate as EGD for diagnosing mucosal pathology and takes approximately 1 minute longer.(1; 2) Previously published work by our group suggests that EUS may reduce resource consumption in patients with unexplained abdominal pain.(3) The investigators also showed that refractory dyspepsia with normal EGD and CT, EUS identified signs of occult chronic pancreatitis in up to 20% of cases.(4) More recently, EUS was found to identify previously undiagnosed, potential causes of unexplained abdominal pain in up to 9% of patients, or at least provides the same, if not more information and EGD and abdominal US alone.(2; 5; 6) There are no previous studies that have prospectively compared the yield of EGD and PEUS in emergency room patients. The investigators hypothesize that adding EUS to EGD ("primary EUS" [PEUS]) can safely and more efficiently diagnose or exclude significant gastro-intestinal and pancreatico-biliary pathology in emergency room patients in whom EGD has been requested. The investigators therefore propose a prospective pilot study to determine whether PEUS can reduce LOS and resource utilisation in emergency room patients referred for EGD.

AIM To perform a pilot study to determine whether PEUS reduces emergency room LOS and resource utilisation in emergency room patients referred for EGD.

METHODS

Study design This is an open-label two-arm, single center, superiority trial with 1:1 allocation ratio between EUS and standard intervention EGD.

Site

This study will be performed at the St Luc site of CHUM. Approximately 5000 EGD procedures and 3000 EUS procedures are performed at this site annually. Therefore, there should be sufficient eligible patients for efficient patient recruitment.

Research team A research team composed of the PI, one research nurse, and a biostatistician will coordinate the trial. The research assistant will be responsible for all data collection and patient recruitment (including consent). Statistical analysis will be provided by the biostatistical platform of the CR-CHUM under the supervision of Dr Martin Ladouceur.

Funding There is no external funding for this study.

Patient selection All patients referred for GI consultation in the emergency room at CHUM, site St Luc, are eligible.

Inclusion Criteria EGD requested by the consulting gastroenterologist Informed consent

Exclusion criteria Evidence of hemodynamic instability and/or ongoing active GI bleeding. Any suspicion of obstruction distal to the angle of Treitz. EGD or EUS cannot be performed before 12PM. Previous barium study, EGD, US, abdomino-pelvic CT, or abdomino-pelvic MRI within the last 6 months.

After the EGD request form is received in the GI department, the patient will be transported as usual to the endoscopy unit. Before entering an endoscopy suite, a single research assistant will present the patients the study protocol. After informed consent, each group will be randomized by sealed envelop to EGD or to PEUS. A gastroenterologist other than the one who requested EGD will perform EGD or EUS. Written EGD and PEUS reports will be presented in the standard fashion.

EGD and EUS are both available every day, before 12PM. They will be performed and interpreted by experienced operators (not fellows).

OUTCOMES

Patients in whom EGD is scheduled after GI consultation will be stratified in to 2 groups:

1. abdominal pain syndromes (defined as any pain or discomfort considered to be possibly of GI origin)
2. all other indications.

Primary outcome The primary outcome will be "time to GI diagnosis" (with T0 starting immediately after the procedure report is read and signed by the referring physician). A "GI diagnosis" is defined as diagnosis or confirmation of any condition sufficient to start treatment or to modify the existing therapeutic regimen.

Secondary outcomes

Secondary outcomes will be:

frequency of conversion to the alternate procedure (EGD to EUS, or EUS to EGD) number of subsequent imaging procedures other than endoscopy complications (defined as any event that prolongs hospital stay)

SAMPLE SIZE CALCULATIONS Given the novelty of the primary outcome of this study ("time to diagnosis, discharge, or admission"), there are no reliable data on which a sample-size estimate can be calculated. The investigators propose a pilot approach, with 40 patients per randomisation group (80 patients in total). This would be followed by an analysis to further clarify the appropriate sample size.

4.4 Expected Duration of Study Given our current patient volumes, the investigatorsshould be able to recruit 1 person per day (5 per week). This should require approximately 16 weeks (4 months) to complete this pilot project. Given that the primary endpoint is likely to occur in less than 3-4 days, the entire study duration until complete follow of the last patient would be approximately 17 weeks. To be conservative, and allow for unexpected contingencies, we propose an estimate for pilot study duration of 8 months.

ELIGIBILITY:
Inclusion Criteria:

* EGD requested by the consulting gastroenterologist
* Informed consent

Exclusion Criteria

* Evidence of hemodynamic instability and/or ongoing active GI bleeding.
* Any suspicion of obstruction distal to the angle of Treitz.
* EGD or EUS cannot be performed before 12PM.
* Previous barium study, EGD, US, abdomino-pelvic CT, or abdomino-pelvic MRI within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
time to GI diagnosis | 1 day
  The primary outcome will be "time to GI diagnosis" (with T0 starting immediately after the procedure report is read and signed by the referring physician). A "GI diagnosis" is defined as diagnosis or confirmation of any condition sufficient to start treatment or to modify the existing therapeutic regimen.

SECONDARY OUTCOMES:
frequency of conversion to the alternate procedure (EGD to EUS, or EUS to EGD) | 1 day
  Number of subjects who were sent to do the alternate procedure
number of subsequent imaging procedures other than endoscopy | 1 day
  Includes scans, ultrasounds, MRI, etc.
Complications | 1 day
  Defined as any event that prolongs hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Anand Sahai, M.D, Principal Investigator — CRCHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haider S, Kahaleh M. The use of endoscopic clipping devices in the treatment of iatrogenic duodenal perforation. Gastroenterol Hepatol (N Y). 2010 Oct;6(10):660-1. No abstract available. PMID 21103446
- [Background] Chang KJ, Erickson RA, Chak A, Lightdale C, Chen YK, Binmoeller KF, Albers GC, Chen WP, McLaren CE, Sivak MV, Lee JG, Isenberg GA, Wong RC. EUS compared with endoscopy plus transabdominal US in the initial diagnostic evaluation of patients with upper abdominal pain. Gastrointest Endosc. 2010 Nov;72(5):967-74. doi: 10.1016/j.gie.2010.04.007. Epub 2010 Jul 22. PMID 20650452
- [Background] Sahai AV, Penman ID, Mishra G, Williams D, Pearson A, Wallace MB, van Velse A, Hoffman BJ, Hawes RH. An assessment of the potential value of endoscopic ultrasound as a cost-minimizing tool in dyspeptic patients with persistent symptoms. Endoscopy. 2001 Aug;33(8):662-7. doi: 10.1055/s-2001-16223. PMID 11490381
- [Background] Sahai AV, Mishra G, Penman ID, Williams D, Wallace MB, Hadzijahic N, Pearson A, Vanvelse A, Hoffman BJ, Hawes RH. EUS to detect evidence of pancreatic disease in patients with persistent or nonspecific dyspepsia. Gastrointest Endosc. 2000 Aug;52(2):153-9. doi: 10.1067/mge.2000.107910. PMID 10922084
- [Background] Thompson MB, Ramirez JC, De La Rosa LM, Wood AS, Desai S, Arjunan A, Song J, Erickson RA. Endoscopic ultrasound in the evaluation of chronic upper abdominal pain of unknown etiology: a retrospective chart review examining the efficacy of EUS in determining a new diagnosis. J Clin Gastroenterol. 2015 Feb;49(2):e17-20. doi: 10.1097/MCG.0000000000000174. PMID 25569224
- [Background] Attasaranya S, Ovartlarnporn B. The possible diagnostic role of endoscopic ultrasound in patients with dyspepsia. J Med Assoc Thai. 2005 Nov;88(11):1660-5. PMID 16471116